CLINICAL TRIAL: NCT01965483
Title: Weekly Hypofractionated Radiotherapy in Breast Cancer: a Phase 2 Clinical Trial
Brief Title: Phase 2 Study of Adjuvant Radiotherapy in Breast Cancer Using a Once a Week Hypofractionated Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Ceara (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 009/2013
Record Dates: First submitted 2013-10-13; First posted 2013-10-18 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Breast Neoplasms
Keywords: radiotherapy; adjuvant; weekly hypofractionation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: ONCE-WEEKLY HYPOFRACTIONATED RADIOTHERAPY FOR BREAST CANCER:
  PHASE II NON-RANDOMIZED CLINICAL TRIAL
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weekly radiation (Experimental): once-weekly breast irradiation
  Interventions: Radiation: once-weekly breast irradiation

INTERVENTIONS:
Radiation: once-weekly breast irradiation

SUMMARY:
The implementation of a weekly hypofractionated radiation could be an advantageous alternative. The convenience of less treatment days could cause a greater adherence, decrease of costs and increase the offer of radiotherapy to major number of patients in underserved areas.

The purpose of this study is to determine in women with diagnosis of initial breast cancer undergoing breast-conserving surgery the effects of the adjuvant radiotherapy using a once a week regimen, with 5 fractions in total. The study will analyze the acute toxicity of radiation, the patient's self referred quality of life, the cosmetic breast appearance, as well the oncological safety. It will also be analyzed the viability of this more contracted regimen in our community setting, regarding the patient's adherence to the treatment.

DETAILED DESCRIPTION:
The patients will be told about the study and have all their questions clarified. After agreeing to participate in the study they must sign a declaration of free and informed consent.

All the radiation treatments will be carried out in the Radiotherapy Department of the Haroldo Juacaba Hospital. The primary intention of the radiotherapy (RT) is to treat the entire breast. Initially, with the patient in supine position and the making of an individual immobilization device, it will be done a pre-planning in a conventional radiotherapy simulator. After that, a CT-scan will be performed for the three-dimensional conformal radiation planning.

The contouring of the treatments volumes (target volumes and organs-at-risk) and the dosimetric calculations will be performed in the Eclipse treatment planning system (Varian Medical Systems, Palo Alto-CA, USA). The total dose prescribed will be of 30 Gy, in 5 fractions of 6.0 Gy, 1 fraction per week, 1 week apart in the same weekday. In the dosimetric analysis, at least 95% of the breast target-volume must be covered by ≥ 95% of the prescription dose. The point of maximum dose must be less than 110%.

Clinical evaluations will be carried out weekly during the treatment course and in the 4th and 8th weeks after the conclusion of RT. The toxicity will be graduated according to the Common Toxicity Criteria for Adverse Events (CTCAE), v 3.0.

Breast photographs will be held initially and 6 and 12 months after treatment. Breast cosmetic appearance will evaluated by 2 radiation oncologists and classified according to the Harvard scale. The patient's self-referred quality-of-life (QoL) data will be collected in 3 different moments, before the begging of RT just at the end and 1 month after the conclusion of RT. The QoL evaluation tools to be used are the European Organization for Research and Treatment of Cancer (EORTC) QLQ-30 and the breast cancer specific module QLQ-BR23 questionnaires. The projected sample size is 40 patients.

Which patient has the right of no longer be part of the study at any time, if this will be her desire. The study will be interrupted in the case of severe toxicity (≥ grade IV), death caused by the treatment and/or local recurrence superior than the expected, as the reported by literature. Interim analyzes will be performed every 6 months for better monitoring of these possible outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Breast carcinoma
* Submitted to breast conserving surgery with pos-op free margins status
* Early stage: pT1-2N0

Exclusion Criteria:

* Positive pathological margins
* Submitted to chemotherapy, either neoadjuvant or adjuvant
* Previous breast reconstruction
* Bilateral breast cancer
* Previous thoracic irradiation
* Collagen disease

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number patients with adverse events | RT duration, 5 weeks

SECONDARY OUTCOMES:
Cosmetic appearance | One year
Number of local failures after RT | One year
Cancer specific survival | One year
Quality-of-life | one month
Adherence to RT regimen | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Conceicao Souza, MD, PhD, Principal Investigator — Instituto do Cancer do Ceara
Locations (1):
- Radiotherapy Department, Instituto do Cancer do Ceara, Fortaleza, Ceará, Brazil

REFERENCES:
- [Background] FAST Trialists group; Agrawal RK, Alhasso A, Barrett-Lee PJ, Bliss JM, Bliss P, Bloomfield D, Bowen J, Brunt AM, Donovan E, Emson M, Goodman A, Harnett A, Haviland JS, Kaggwa R, Morden JP, Robinson A, Simmons S, Stewart A, Sydenham MA, Syndikus I, Tremlett J, Tsang Y, Wheatley D, Venables K, Yarnold JR. First results of the randomised UK FAST Trial of radiotherapy hypofractionation for treatment of early breast cancer (CRUKE/04/015). Radiother Oncol. 2011 Jul;100(1):93-100. doi: 10.1016/j.radonc.2011.06.026. PMID 21752481
- [Background] Dragun AE, Quillo AR, Riley EC, Roberts TL, Hunter AM, Rai SN, Callender GG, Jain D, McMasters KM, Spanos WJ. A phase 2 trial of once-weekly hypofractionated breast irradiation: first report of acute toxicity, feasibility, and patient satisfaction. Int J Radiat Oncol Biol Phys. 2013 Mar 1;85(3):e123-8. doi: 10.1016/j.ijrobp.2012.10.021. Epub 2012 Nov 27. PMID 23195779
- [Background] Kirova YM, Campana F, Savignoni A, Laki F, Muresan M, Dendale R, Bollet MA, Salmon RJ, Fourquet A; Institut Curie Breast Cancer Study Group. Breast-conserving treatment in the elderly: long-term results of adjuvant hypofractionated and normofractionated radiotherapy. Int J Radiat Oncol Biol Phys. 2009 Sep 1;75(1):76-81. doi: 10.1016/j.ijrobp.2008.11.005. Epub 2009 Jan 23. PMID 19168297
- [Derived] Reboucas LM, Campos CS, D'Amico GM, Lustosa AB, Fregnani JH. Once-weekly hypofractionated radiotherapy for breast cancer: First results of a phase II clinical trial. Breast J. 2019 Sep;25(5):953-957. doi: 10.1111/tbj.13372. Epub 2019 Jun 4. PMID 31165541